CLINICAL TRIAL: NCT05936281
Title: A Randomized, Open-lable, Multi-center, Active-controlled Phase 2 Study for Evaluating Efficacy and Safety of Genakumab in Prevention of Acute Flares in Gout Patients Initiating Urate-lowering TherapyUrate-lowering
Brief Title: A Study of the Efficacy of Genakumab in Prevention of Acute Flares in Gout Patients Initiating Urate-lowering TherapyUrate-lowering (GenSci048-202)
Acronym: Gensci 048-202
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 048-202
Record Dates: First submitted 2023-06-30; First posted 2023-07-07 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Gout; Gout Initiating Urate-loweringUrate-lowering Therapy
Keywords: Gout; urate-loweringUrate-lowering therapy
MeSH Terms: conditions — Gout | interventions — Injections; Colchicine

STUDY DESIGN:
Intervention Model Description: Gout patients initiating urate-lowering therapy Group A: Genakumab 100mg single injection; Group B: Genakumab 200mg single injection;Group C: Oral colchicine 0.5mg once a day for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genakumab group (Experimental): Genakumab 100mg single injection、Genakumab 200mg single injection
  Interventions: Drug: Genakumab for injection
- Colchicine group (Active Comparator): Oral colchicine 0.5mg once a day for 12 weeks
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Genakumab for injection — 150 mg/1ml/ vial
  Arms: Genakumab group
Drug: Colchicine — 0.5 mg/table
  Arms: Colchicine group

SUMMARY:
To evaluate the safety and efficacy of Genakumab in prevention of acute flares in gout patients initiating urate-lowering therapyurate-lowering

DETAILED DESCRIPTION:
A randomized, open-lable, multi-center, active-controlled Phase 2 study. Patients are randomized to Genakumab 100mg single injection group, Genakumab 200mg single injection group or oral colchicine 0.5mg once a day.for 12 weeks group.

ELIGIBILITY:
1. Signed written informed consent before any study procedure is performed.
2. Male or female, 18 years ≤ age ≤ 75 years.
3. BMI ≤ 40kg/m2.
4. Confirmed diagnosis of gout meeting the American College of Rheumatology (ACR) 2015 preliminary criteria for the classification of arthritis of primary gout.
5. History of ≥2 gout flare within 12 months prior to screening.
6. Willingness to initiate urate-lowering therapy or having initiated urate-lowering therapy within 1 week prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Mean Number of Gout Flares Per Participant | Baseline to Week 12

SECONDARY OUTCOMES:
Proportion of Participants With at Least 1 Gout Flare Within 12 Weeks After Randomization | Baseline to Week 12
Time from Randomization to the First Flare | Baseline to Week 12
Mean duration of flares | Baseline to Week 12
5. Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) | Baseline to Week 12

OTHER OUTCOMES:
6. Immunogenic Outcome The incidence of anti-drug antibodies and the incidence of neutralizing antibody | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Hejian Zou, Principal Investigator — Fudan University Affiliated Huashan Hospital
Locations (1):
- Fudan University Affiliated Huashan Hospital, Shanghai, Shanghai Municipality, China